CLINICAL TRIAL: NCT01138670
Title: Complications Following Pacemaker or ICD Implantation in Denmark
Brief Title: Complications Following Pacemaker or Implantable Defibrillator Cardioverter (ICD) Implantation in Denmark
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: SKS-REK-2
Record Dates: First submitted 2010-05-25; First posted 2010-06-07 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Pacemaker; Defibrillators, Implantable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac device group

SUMMARY:
This study examines possible risk factors with regard to complications following pacemaker or implantable defibrillator cardioverter (ICD) implantation.

DETAILED DESCRIPTION:
This study examines possible risk factors with regard to complications following pacemaker or implantable defibrillator cardioverter (ICD)implantation. Furthermore validation af the Danish Pacemaker and ICD Register will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving a cardiac device (pacemaker, cardiac resynchronization therapy (CRT) or implantable defibrillator cardioverter (ICD)), or undergoing a reoperation

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Danish patients receiving a cardiac device (pacemaker, cardiac resynchronization therapy (CRT) or implantable defibrillator cardioverter (ICD)), or undergoing a reoperation from May 2010 to April 2011.
Sampling Method: Probability Sample
Enrollment: 5500 (Estimated)
Dates: Start 2010-05; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
complication rate | 3 months
  any complication that require treatment There is no 'Safety and Tolerability' or 'Pain' measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Rikke E Kirkfeldt, MD, Principal Investigator — Aarhus Universitetshospital, Skejby
Locations (1):
- Aarhus Universitetshospital, Skejby, Aarhus, Denmark